CLINICAL TRIAL: NCT04620447
Title: Development of Intelligent Virtual Reality Therapy System (IVRTS) and Testing Its Clinical Efficacy: Revolutionizing Evidence-Based Psychotherapy
Brief Title: Intelligent Virtual Reality Therapy System and Testing Its Clinical Efficacy
Acronym: IVRTS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College of Medical Sciences, India (Individual)
Collaborators: Norwegian University of Science and Technology (Other); Indraprastha Institute of Information Technology Delhi (Other)
Responsible Party: Principal Investigator, Akshay Kumar, Assistant Professor and Clinical Consultant, University College of Medical Sciences, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/1/333011/HRD
Record Dates: First submitted 2020-10-20; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Phobias; Acrophobia; Anxiety
Keywords: Anxiety; Virtual Reality; Phobias; Clinical Intervention
MeSH Terms: conditions — Phobic Disorders; Acrophobia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: To achieve the stated objective, a two-fold approach comprising of qualitative and quantitative analysis was undertaken. A 7-week intervention course was designed for each subject to reduce symptoms and enhance quality of life as well as to establish clinical efficacy. .
  The participants were assigned to three groups using circumstantial sampling methodology. Group 1: IVRTS, Group 2: Mindfulness, Group 3: Cognitive Behavior Therapy, Group 4: Control Group.
  Further study carried out A-B-A research design (Pre and Post intervention) which mainly involved establishing a baseline condition, introducing an experimental treatment and then returning to the baseline. The subjects completed standardized self-report measures of Hamilton Anxiety Inventory (HAM-A), Subjective Units of Dysfunction (SUDS) and WHO Quality of Life - BREF Questionnaire (QOL-BREF) at baseline, after seven intervention sessions post assessments on the same scales were repeated to assess the efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness Meditation (Active Comparator): A 7-week intervention course was designed for each subject to reduce symptoms and enhance quality of life as well as to establish clinical efficacy.
  Number of Participants: 125
  Dropouts: 7
  Final number of participants: 118
  Mindfulness Meditation intervention was conducted on a sample of 118 patients diagnosed with Acrophobia co-morbid with generalized anxiety who underwent the intervention at The University College of Medical Sciences and GTB hospital.
  study carried out A-B-A research design which mainly involved establishing a baseline condition, introducing an experimental treatment and then returning to the baseline. The subjects completed standardized self-report measures of Hamilton Anxiety Inventory (HAM-A), Subjective Units of Dysfunction (SUDS) and WHO Quality of Life - BREF Questionnaire (QOL-BREF) at baseline, after seven intervention sessions post assessments on the same scales were repeated to assess the efficacy.
  Interventions: Other: Intelligent Virtual Reality Therapy System (IVRTS)
- Cognitive Behavior Therapy (Active Comparator): A 7-week intervention course was designed for each subject to reduce symptoms and enhance quality of life as well as to establish clinical efficacy.
  Number of Participants: 125
  Dropouts: 19
  Final number of participants: 102
  Cognitive Behavior Therapy intervention was conducted on a sample of 118 patients diagnosed with Acrophobia co-morbid with generalized anxiety who underwent the intervention at The University College of Medical Sciences and GTB hospital.
  study carried out A-B-A research design which mainly involved establishing a baseline condition, introducing an experimental treatment and then returning to the baseline. The subjects completed standardized self-report measures of Hamilton Anxiety Inventory (HAM-A), Subjective Units of Dysfunction (SUDS) and WHO Quality of Life - BREF Questionnaire (QOL-BREF) at baseline, after seven intervention sessions post assessments on the same scales were repeated to assess the efficacy.
  Interventions: Other: Intelligent Virtual Reality Therapy System (IVRTS)
- Novel 'Intelligent Virtual Reality Therapy System' (IVRTS) (Active Comparator): A 7-week intervention course was designed for each subject to reduce symptoms and enhance quality of life as well as to establish clinical efficacy.
  Number of Participants: 125
  Dropouts: 10
  Final number of participants: 115
  Novel 'Intelligent Virtual Reality Therapy System' (IVRTS) was conducted on a sample of 118 patients diagnosed with Acrophobia co-morbid with generalized anxiety who underwent the intervention at The University College of Medical Sciences and GTB hospital.
  study carried out A-B-A research design which mainly involved establishing a baseline condition, introducing an experimental treatment and then returning to the baseline. The subjects completed standardized self-report measures of Hamilton Anxiety Inventory (HAM-A), Subjective Units of Dysfunction (SUDS) and WHO Quality of Life - BREF Questionnaire (QOL-BREF) at baseline, after seven intervention sessions post assessments on the same scales were repeated to assess the efficacy.
  Interventions: Other: Intelligent Virtual Reality Therapy System (IVRTS)
- Control Group (No Intervention): A 7-week intervention course (In this case, no intervention) was designed for each subject to reduce symptoms and enhance quality of life as well as to establish clinical efficacy.
  Number of Participants: 125
  Dropouts: 0
  Final number of participants: 125
  study carried out A-B-A research design which mainly involved establishing a baseline condition, introducing an experimental treatment and then returning to the baseline. The subjects completed standardized self-report measures of Hamilton Anxiety Inventory (HAM-A), Subjective Units of Dysfunction (SUDS) and WHO Quality of Life - BREF Questionnaire (QOL-BREF) at baseline, after seven intervention sessions post assessments on the same scales were repeated to assess the efficacy.

INTERVENTIONS:
Other: Intelligent Virtual Reality Therapy System (IVRTS) — The approach of the Novel Intelligent Software interface approaches follows the basic premise that human beings think in terms of images rather than words. While the existing modes of treatment for phobias rely mainly on talk therapies and counseling; This novel intelligent software treatment methodology deals with the development of VR programs integrated with hardware for simulating various phobia-inducing situations, followed by novel automated integrated most effective psychotherapy; altering these images to reduce the anxiety experienced. Our treatment package includes a VR device integrated with easily comprehensible voice commands, along with a user manual and easy user interface, thereby reducing the effort of training required for operating the device. The framework is a combination of the therapy methodologies with VR, motion sensors and biofeedback.
  Arms: Cognitive Behavior Therapy; Mindfulness Meditation; Novel 'Intelligent Virtual Reality Therapy System' (IVRTS)

SUMMARY:
Objective: To take the existing VR technology to the next level, the investigators developed a novel Intelligent Virtual Reality Therapy System (IVRTS). The objective of this project had three aspects: Namely, development of the novel IVRTS technology involving the development of a hardware device, development of Artificially Intelligent Psychotherapeutic software-interface and testing it's clinical efficacy. Methods: It used a two-phased methodology; Development of the novel technology and testing its Clinical Efficacy. After development of Novel IVRTS. A 7-week intervention was designed for each subject. The sample of 500 patients, meeting the criteria of Acrophobia and Anxiety, underwent the interventions at The GTB hospital (The University of Delhi), for a total 3500 sessions, ranging 5250 hours for over 2 years. The subjects were randomly divided into 4 groups: IVRTS Group, Mindfulness group, CBT group and Control Group. The ethics committee and clinical trial registration number is 33011. Development of this technology would be a land-mark innovation.

DETAILED DESCRIPTION:
Many researchers have proved the usefulness of Virtual Reality Technology in the treatment of Psychological Disorders, and many studies have quoted efficacy of the treatment as well. The research in the VR field is progressing but still is at a very nascent stage10. However, despite some VR projects being worked upon in the current times, the technology is not being used widely, due to its limited proven efficacy. The current VR technology that exists is only limited to placing a patient in his or her phobic situation virtually and not beyond that. In this current project the investigators attempted to fill this gap by using two important novel technological developments. Firstly, the investigators moved beyond just the visual imaging and added haptic touch sensors as well as motion sensors to the device. Secondly, the investigators developed an automated intelligent interactive Psychotherapy software to compliment the virtual reality as a part of the device and finally the investigators tested its clinical efficacy to make sure the novel technology is effective. When the world is sitting on the verge of a Mental Health Crisis due to the global pandemic. The investigators need to revolutionize the Psychotherapy modality for two reasons, first being, the shortage of Mental Health Professionals compared the anticipated cases that would need help due to this unique global condition and secondly accessibility. When social isolation has become the norm for prevention, one needs innovative tools to be able to effectively handle the situation sitting at home, and yet be equally effective, if not more. This is the dire need of the society today and the project has immense potential as well has huge social impact for the treatment of Anxiety Disorders which currently effects 80% of the world population according to the World Health Organization, which is predicted to grow further due to the current global pandemic. The development of this novel technology would reduce the cost of treatment of Anxiety disorders, PTSD and Phobias considerably, which would make interventions viable for people across the world currently not being able to afford long term Psychological sessions. It would also reduce the treatment time by approximately half. It would make the accessibility of treatment widely available and more comfortable for the masses.

The current Virtual Reality technology to treat Anxiety phobias and general stress was at a very nascent stage, where a subject was immersed into phobic situation and is expected to get stage-wise comfortable with it. The current existing Virtual Reality technology to treat phobia is still relatively new and lacks both theoretical and clinical research. VR applications need to go beyond only immersing the person into a phobic situation. This proposed research & development project aimed to integrate complex and proven effective psychotherapies (visual, auditory, interactive, kinesthetic, motion sensing and tactile), automated, intelligent and integrated with the Virtual Reality Technology, which the subject or patient will be able to control and undergo themselves, then it's initial clinical efficacy was examined. Keller and Bunnel explain, Virtual Reality being a technological system helps subjects to experience computer and machine generated situations in lab settings. The technology is being widely utilized in Psychological treatment and research. Rizzo, mentions that people totally experience Virtual reality when it mimics real life at the highest possible level and the users start believing that the situation simulates the real actual world experience that it is recreating. This project developed new technology, devices, and intelligent psychotherapeutic software programs in VR for curing phobias, anxiety, stress and even stress management. The current technology in this field that existed is only at a level of immersing a subject in a realistic VR image/scene and is not beyond that. Currently, this technology was not useful in the treatment, and that is the reason had not entered widely in clinical settings yet.

To take this technology to the next level, one needed to develop a novel VR technology/device, which is intelligent, as well as which would interact and stimulate "Whole brain activation" and help the subject overcome phobia/stress/anxiety effectively. This required developing a device which had motion sensors, interactive sensors which allowed the subject to feel and interact with the image, scenario, program real- time and other psychotherapeutic intelligent technological hardware components and intelligent interactive psychotherapeutic software programs fostering this process, all built in one integrated compact device.

Furthermore, the main components of this project included -Hardware, software, system interfaces and data. The data being collected by the wireless sensor contains information about the health status of the user is stored in a database. Health status data included information about blood pressure, heart rate and other physiological parameters as well.

This project is aimed to develop both hardware and software technology and finally test its clinical efficacy to treat Phobias, General Anxiety, Stress and PTSD. According to the DSM 5 published by the American Psychiatry Association, specific phobias are associated with fear or Anxiety attached to a specific situation or Object Like water, animals, animals, public speaking, needles, heights, blood etc. DSM Also defines Generalized anxiety disorder (GAD) as a condition in which a person Feels intrusive, excessive, and persistent worrying to the extent that daily functioning becomes difficult.

Anxiety and Stress is becoming a global epidemic, The World Health Organization, estimates that 1 in 3 from Clinical Anxiety and 1 in 5 individuals are suffering from Clinical Depression. About 80% of the world is suffering from general stress.

It is said that situation improves with pumping in of resources and putting in efforts; but in this situation despite putting in huge funds, highest quality of resources, the best human minds and fierce efforts, the problem is only increasing. The development of this novel technology will be a landmark step towards the intervention of these conditions the world is battling in present times.

NOVELTY OF THE PROJECT

The approach of the Novel Intelligent Software interface approaches follows the basic premise that human beings think in terms of images rather than words. While the existing modes of treatment for phobias rely mainly on talk therapies and counseling; This novel intelligent software treatment methodology deals with the development of VR programs integrated with hardware for simulating various phobia-inducing situations, followed by novel automated integrated most effective psychotherapy; altering these images to reduce the anxiety experienced. Our treatment package includes a VR device integrated with easily comprehensible voice commands, along with a user manual and easy user interface, thereby reducing the effort of training required for operating the device. The framework is a combination of the therapy methodologies with VR, motion sensors, biofeedback and fNIRS. This would eliminate the need for a therapist by making the patient self-sufficient in handling the overall treatment themselves. In the long run, this would prove to be more cost-effective and socially accessible.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting the Psychiatry OPD of University College of Medical Sciences of the University of Delhi and the attached GTB Hospital.
* Patients who reported fear of heights and scored mild, moderate and Severe anxiety as assessed on Hamilton Anxiety Inventory.
* The patients in age group between 18 to 60 years of age.

Exclusion Criteria:

* Patients who had any Psychotic disorder were not selected for the study.
* Patients who had co-morbidity with any Psychiatry or medical illness other than Acrophobia and Anxiety were not selected for the study.
* Patients below 18 years of age and over 60 years of age were not selected for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in of symptom intensity of acrophobia in the Intelligent Virtual Reality Therapy System Group as compared to Mindfulness Meditation and Cognitive Behavior Therapy Groups. As assessed on Hamilton Anxiety Inventory. | 7 weeks
  Change in symptom intensity as assessed on Hamilton Anxiety Inventory. With lower score indicating higher effectiveness. 0 Being the lowest score and 56 being the highest.
Change in symptom intensity of acrophobia in the Intelligent Virtual Reality Therapy System Group as compared to Mindfulness Meditation and Cognitive Behavior Therapy Groups. As assessed on Subjective Units of Dysfunction Scale. | 7 weeks
  Change in symptom intensity of symptoms as assessed on Subjective Units of Dysfunction Scale. With lower score indicating higher effectiveness. 0 being the lowest score and 5 being the highest.
Change in symptom intensity of acrophobia in the Intelligent Virtual Reality Therapy System Group as compared to Cognitive Behavior Therapy Group and Cognitive Behavior Therapy Groups. As assessed on World Health Organization Quality of Life Bref | 7 weeks
  Change in symptom intensity level of Well-being as assessed on World Health Organization Quality of Life Bref Scale. Higher the score more the well-being levels. 26 being the lowest score and 120 being the highest score.
Change in symptom intensity of acrophobia Pre and Post Intervention in Intelligent Virtual Reality Therapy System as compared to the Control Group. As assessed on Hamilton Anxiety Inventory. | 7 weeks
  Change in symptom intensity of symptoms as assessed on Hamilton Anxiety Inventory. With lower score indicating higher effectiveness. 0 Being the lowest score and 56 being the highest.
Change in symptom intensity of acrophobia Pre and Post Intervention in Intelligent Virtual Reality Therapy System as compared to the Control Group. As assessed on The Subjective Units of Dysfunction Scale. | 7 weeks
  Reduction of symptoms as assessed on Subjective Units of Dysfunction Scale. With lower score indicating higher effectiveness. 0 being the lowest score and 5 being the highest.
Change in symptom intensity of acrophobia Pre and Post Intervention in Intelligent Virtual Reality Therapy System as compared to the Control Group. As assessed on World Health Organization Quality of Life - BREF | 7 weeks
  Enhanced well-being as assessed on World Health Organization Quality of Life Bref Scale. Higher the score, better the well-being levels. Higher the score more the well-being levels. 26 being the lowest score and 120 being the highest score.

CONTACTS AND LOCATIONS:
Overall Officials: Manjit Singh Bhatia, MBBS; MD, Study Director — University College Of Medical Sciences (UCMS) And GTB Hospital
Locations (1):
- University College of Medical Sciences (UCMS) and GTB Hospital, Department of Psychiatry, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Committee on Developing Evidence-Based Standards for Psychosocial Interventions for Mental Disorders; Board on Health Sciences Policy; Institute of Medicine; England MJ, Butler AS, Gonzalez ML, editors. Psychosocial Interventions for Mental and Substance Use Disorders: A Framework for Establishing Evidence-Based Standards. Washington (DC): National Academies Press (US); 2015 Sep 18. Available from http://www.ncbi.nlm.nih.gov/books/NBK305126/ PMID 26203478
- [Result] Cartreine JA, Ahern DK, Locke SE. A roadmap to computer-based psychotherapy in the United States. Harv Rev Psychiatry. 2010 Mar-Apr;18(2):80-95. doi: 10.3109/10673221003707702. PMID 20235773
- [Result] Barnett JE. Utilizing technological innovations to enhance psychotherapy supervision, training, and outcomes. Psychotherapy (Chic). 2011 Jun;48(2):103-8. doi: 10.1037/a0023381. PMID 21639653
- [Result] Fairburn CG, Cooper Z. Therapist competence, therapy quality, and therapist training. Behav Res Ther. 2011 Jun;49(6-7):373-8. doi: 10.1016/j.brat.2011.03.005. Epub 2011 Mar 21. PMID 21492829
- [Result] Kobak KA, Craske MG, Rose RD, Wolitsky-Taylor K. Web-based therapist training on cognitive behavior therapy for anxiety disorders: a pilot study. Psychotherapy (Chic). 2013 Jun;50(2):235-47. doi: 10.1037/a0030568. Epub 2013 Feb 11. PMID 23398031
- [Result] Freeman D, Lister R, Waite F, Yu LM, Slater M, Dunn G, Clark D. Automated psychological therapy using virtual reality (VR) for patients with persecutory delusions: study protocol for a single-blind parallel-group randomised controlled trial (THRIVE). Trials. 2019 Jan 29;20(1):87. doi: 10.1186/s13063-019-3198-6. PMID 30696471
- [Result] Freeman D, Haselton P, Freeman J, Spanlang B, Kishore S, Albery E, Denne M, Brown P, Slater M, Nickless A. Automated psychological therapy using immersive virtual reality for treatment of fear of heights: a single-blind, parallel-group, randomised controlled trial. Lancet Psychiatry. 2018 Aug;5(8):625-632. doi: 10.1016/S2215-0366(18)30226-8. Epub 2018 Jul 11. PMID 30007519
- [Result] Maples-Keller JL, Bunnell BE, Kim SJ, Rothbaum BO. The Use of Virtual Reality Technology in the Treatment of Anxiety and Other Psychiatric Disorders. Harv Rev Psychiatry. 2017 May/Jun;25(3):103-113. doi: 10.1097/HRP.0000000000000138. PMID 28475502
- [Result] Garcia-Palacios A, Hoffman H, Carlin A, Furness TA 3rd, Botella C. Virtual reality in the treatment of spider phobia: a controlled study. Behav Res Ther. 2002 Sep;40(9):983-93. doi: 10.1016/s0005-7967(01)00068-7. PMID 12296495
- [Result] Miloff A, Lindner P, Hamilton W, Reuterskiold L, Andersson G, Carlbring P. Single-session gamified virtual reality exposure therapy for spider phobia vs. traditional exposure therapy: study protocol for a randomized controlled non-inferiority trial. Trials. 2016 Feb 2;17:60. doi: 10.1186/s13063-016-1171-1. PMID 26833396

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT04620447/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT04620447/ICF_001.pdf